CLINICAL TRIAL: NCT01454882
Title: Measuring Free-living Energy Expenditure Using Direct Calorimetry
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Alabama at Birmingham (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 11-1324; R01DK091287 (NIH)
Record Dates: First submitted 2011-10-14; First posted 2011-10-19 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Temperature; Clothing; Sex; Age; Adiposity
Keywords: Direct calorimetry; Indirect calorimetry; Energy Expenditure
MeSH Terms: conditions — Coitus; Obesity

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Behavioral effects of clothing and temperature: In this first study, we will determine how variations in clothing and ambient temperature influence the accuracy of EE determined from measurements of total heat production. 65 individuals will be studied. This will be a randomized cross-over trial with two within subject factors: 1) ambient temperature and 2) amount of clothing. There will be two temperature conditions; warm temperature [WT, 75°F (24°C)] and cool temperature [CT, 60°F (16°C)]. During each condition, subjects will vary the amount of clothing they are wearing at specified times
  Interventions: Behavioral: Effects of Clothing; Behavioral: Effects of Temperature
- Behavioral effects of age, sex, and adiposity: THe aim of this study is to Determine how age, sex, and adiposity influence the accuracy of EE determined from measurements of total heat production . This will be a randomized study with two within subject conditions(high and low physical activity levels). A heterogenous sample of adult men and women in stable health will be studied. We will study subjects across a wide range of weight (up to 300 lbs) and age range (≥ 18 yrs).
  Interventions: Behavioral: Low Physical Activity; Behavioral: High Physical Activity
- Effects of free living energy expenditure: The primary aim of this study is to compare the accuracy of measuring free-living energy expenditure in humans measured using portable direct calorimetry. This will be a comparison study; TDEE will be measured simultaneously for 14 days using direct calorimetry and doubly labeled water. A heterogeneous sample of adult men and women in stable health will be studied. We will study subjects across a wide range of weight (up to 300 lbs) and age (>18 yrs).
  Interventions: Behavioral: Direct calorimetry and doubly labeled water

INTERVENTIONS:
Behavioral: Effects of Clothing — There will be two temperature conditions; warm temperature [WT, 75°F (24°C)] and cool temperature [CT, 60°F (16°C)]. During each condition, subjects will vary the amount of clothing they are wearing at specified times
  Groups: Behavioral effects of clothing and temperature
Behavioral: Effects of Temperature — There will be two temperature conditions; warm temperature [WT, 75°F (24°C)] and cool temperature [CT, 60°F (16°C)]. During each condition, subjects will vary the amount of clothing they are wearing at specified times
  Groups: Behavioral effects of clothing and temperature
Behavioral: Low Physical Activity — This will be a randomized study with two within subject conditions (high and low physical activity levels)
  Groups: Behavioral effects of age, sex, and adiposity
Behavioral: High Physical Activity — This will be a randomized study with two within subject conditions (high and low physical activity levels)
  Groups: Behavioral effects of age, sex, and adiposity
Behavioral: Direct calorimetry and doubly labeled water — TDEE will be measured simultaneously for 14 days using direct calorimetry and doubly labeled water. A heterogeneous sample of adult men and women in stable health will be studied.
  Groups: Effects of free living energy expenditure

SUMMARY:
Although instruments such as pedometers and heart rate monitors are helpful for those who use exercise to maintain their weight, they do not actually measure calories expended, which is a critical piece of information necessary for sustained weight management. The purpose of this study is to determine the accuracy of a new device that measures calories burned based upon heat produced by the body. Since heat production is directly proportional to calories burned, this device has the potential to accurately measure energy expended in many different settings.

DETAILED DESCRIPTION:
Current approaches to measuring total daily energy expenditure (TDEE) in free-living individuals are limited by cost, accuracy, and lack of sensitivity to specific activities. Accurate, reliable, and low cost approaches for measuring TDEE are needed not only to improve clinical outcomes (e.g. weight management), but also to meet public health research objectives. In humans, EE is proportional to total heat loss, which is the sum of conductive, convective, radiant and evaporative heat flows, and measurement of heat loss is the basis of direct calorimetry. However, it has not been possible to accurately measure all forms of heat flux in free-living humans, particularly evaporative heat loss, which can be a substantial component of total heat production. A recently developed heat flow gauge with the capacity to measure all forms of heat flux has shown promise in proof of concept trials and pilot studies, but its accuracy in measuring TDEE has not yet been thoroughly tested. Moreover, how accuracy is affected by factors such as clothing, ambient temperature, and adiposity has not been studied. The objectives of the proposed research are to a) refine the measurement of TDEE based on total heat flux by determining how factors such as clothing, ambient temperature, age, sex, and body composition influence accuracy; b) compare the accuracy of this approach against the criterion measurements of Doubly Labeled Water (DLW) and whole-room indirect calorimetry; and c) compare the accuracy against a similar instrument that measures heat flux, but is not capable of directly measuring the evaporative component. The proposed research is innovative because it will test the accuracy of an approach that is based on a physiological signal (heat production) which is directly proportional to EE. In addition to accurately measuring TDEE, identifying and distinguishing different types of physical activity is an important goal of physical activity related research, but the capacity to do so is limited. Thus, an additional goal of the proposed research is to determine if measurement of changes in heat flux can be used to identify EE in specific bouts of activity and to differentiate between upper body and lower body activity. The proposed studies will permit refinement of a technology that will have major impact in both clinical practice and research. This new approach will potentially provide substantive improvements in the measurement of TDEE in free-living humans and in the assessment of physical activity and the associated energy cost.

ELIGIBILITY:
These studies will be conducted in Denver. CO. Eligible participants will be those local to the University.

Study #1 (Effects of clothing and temperature)

Inclusion Criteria

* Body mass index (BMI) 19-25 kg/m2
* Age 18-45 years

Exclusion criteria

* Self-reported acute or chronic disease (e.g. diabetes, heart disease, thyroid disease)
* Tobacco use (cigarettes, cigars, or chewing tobacco) within the past 6 months
* Females who are or who were recently (past year) pregnant or lactating.
* Resting diastolic blood pressure > 100 mm HG or resting systolic blood pressure > 160 mm HG
* Contra-indications to exercise (e.g. orthopedic limitations)

Study #2 (Effect of age, sex, and adiposity)

Inclusion Criteria • Age ≥18 yrs

Exclusion criteria

* Weight > 300 lbs (due to DXA limitations)
* Self-reported acute or chronic disease (diabetes, heart disease, thyroid disease)
* Tobacco use (cigarettes, cigars, or chewing tobacco) within the past 6 months
* Females who are or who were recently (past year) pregnant or lactating.
* Resting diastolic blood pressure > 100 mm HG or resting systolic blood pressure > 160 mm HG
* Contra-indications to exercise (e.g. orthopedic limitations)

Study #3 (Doubly labeled water)

Inclusion Criteria

• Age ≥18 yrs

Exclusion criteria

* Weight > 300 lbs (due to DXA limitations)
* Self-reported acute or chronic disease (diabetes, heart disease, thyroid disease)
* Tobacco use (cigarettes, cigars, or chewing tobacco) within the past 6 months
* Females who are or who were recently (past year) pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study #1: Lean (body mass index (BMI) < 25.0 kg/m2), adult men and women (18-45 yrs) in stable health will be studied.
  Study #2 & #3: A heterogenous sample of adult men and women in stable health will be studied. We will study subjects across a wide range of weight (up to 300 lbs) and age range (≥ 18 yrs).
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2012-01; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Energy expenditure | 24 hrs to 2 weeks
  The aim of this trial is to determine the accuracy of measuring energy expenditure using portable direct calorimetry. Energy expenditure will be measured with a new device worn on the arm that measures heat flux. The accuracy of the new device will be compared against simultaneous measurements of energy expenditure made using indirect calorimetry and doubly labeled water.

CONTACTS AND LOCATIONS:
Overall Officials: Edward L Melanson, Ph.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver Anschutz Medical Campus, Aurora, Colorado, United States

REFERENCES:
- See also: Screening form — https://redcap.ucdenver.edu/surveys/?s=kxNIBf